CLINICAL TRIAL: NCT02314078
Title: Audit of the Response Time of the Anaesthetic and Surgical Techniques for Crash Caesarean Section
Acronym: Crash
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2013/1043/D
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Pregnancy; Anaesthesia
Keywords: Caesarean section; Emergency; Anaesthesia
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A decision-to-delivery interval of 30 minutes for category-1 Caesarean section deliveries is the standard of practice recommended by clinical guidelines.

DETAILED DESCRIPTION:
Our institution established a protocol for category-1 ('crash') CS to expedite deliveries. This retrospective audit evaluated all women who underwent category-1 CS in KK Women's and Children's Hospital from 2010 to 2013.

ELIGIBILITY:
Inclusion Criteria:

* Category One Caesarean Section at KK Women's and Children's Hospital, Singapore between 2010 to 2013.

Exclusion Criteria:

* No specific exclusion criteria, retrospective audit

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who underwent category one Caesarean section between 2010 to 2013 at KK Women's and Children's Hospital, Singapore.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Decision to delivery interval | 1 hour
  Decision for Caesarean section to delivery of foetus

SECONDARY OUTCOMES:
General anaesthesia | 1 hour
  Rate of general anaesthesia
Neonatal outcome | 1 hour
  APGAR score and cord pH

CONTACTS AND LOCATIONS:
Overall Officials: Ban L Sng, FANZCA, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore